CLINICAL TRIAL: NCT02442349
Title: A Phase II, Open Label, Single-arm Study to Assess the Safety and Efficacy of AZD9291 in Asia Pacific Patients With Locally Advanced/Metastatic Non-Small Cell Lung Cancer Whose Disease Has Progressed With Previous Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy and Whose Tumours Harbour a T790M Mutation Within the Epidermal Growth Factor Receptor Gene.
Brief Title: Phase II Single Arm Study of AZD9291 to Treat NSCLC Patients in Asia Pacific
Acronym: AURA17
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00017
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Phase II, Open Label, Single-arm study, Safety and Efficacy of AZD9291, Asia Pacific, NSCLC with T790M mutation within the Epidermal Growth Factor Receptor Gene
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9291 (Experimental): Once daily tablet 80 mg
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — Once daily tablet 80 mg

SUMMARY:
A Phase II, Open Label, Single-arm Study to Assess the Safety and Efficacy of AZD9291 in Asia Pacific Patients with Locally Advanced/Metastatic Non-Small Cell Lung Cancer whose Disease has Progressed with Previous Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy and whose Tumours harbour a T790M mutation within the Epidermal Growth Factor Receptor Gene

DETAILED DESCRIPTION:
This is a phase II, open label, single arm study assessing the safety and efficacy of AZD9291 (80 mg, orally, once daily) in Asia Pacific patients with a confirmed diagnosis of Epidermal Growth Factor Receptor (EGFR) sensitising mutation positive (ie, G719X, exon 19 deletion, L858R, L861Q) and T790M mutation positive (hereafter referred to as EGFRm+ and T790M+) un-resectable, locally advanced or metastatic NSCLC (Stage IIIB-IV), who have progressed on an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor(EGFR-TKI), either as first line treatment or following one line of EGFR-TKI and one line of platinum containing doublet chemotherapy. Patients must agree to provide a biopsy for central confirmation of T790M mutation status following confirmed disease progression on the most recent treatment regimen. The primary objective of the study is to assess the efficacy of AZD9291 by assessment of Objective Response Rate according to RECIST 1.1 by an Independent Central Review.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years. Patient from Asia Pacific will be enrolled only.
* Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy.
* Radiological documentation of disease progression on the last treatment administered prior to enrolling in the study: following 1st line EGFR TKI treatment but who have not received further treatment OR following prior therapy with an EGFR TKI and a platinum-based doublet chemotherapy. Patients may have also received additional lines of treatment.
* Documented EGFR mutation (at any time since the initial diagnosis of NSCLC) known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q).
* Patients must have central confirmation of tumour T790M mutation positive status from a biopsy sample taken after confirmation of disease progression on the most recent treatment regimen.
* World Health Organisation (WHO) performance status 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
* At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline as ≥10mm in the longest diameter (except lymph nodes which must have short axis ≥15mm) with computerised tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements.
* Females of child-bearing potential using contraception and must have a negative pregnancy test.

Exclusion Criteria:

* Treatment with an EGFR-TKI (eg, erlotinib, gefitinib, icotinib or afatinib) within 8 days or approximately 5x half-life of study entry; any cytotoxic chemotherapy, investigational agents or other anticancer drugs within 14 days of study entry; previous treatment with AZD9291 or a 3rd generation EGFR TKIs; Major surgery within 4 weeks of study entry; radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of study entry; currently receiving treatment with potent inhibitors or inducers of CYP3A4.
* Any unresolved toxicities from prior therapy.
* Unstable spinal cord compression or brain metastases.
* Severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses or infection.
* Refractory nausea and vomiting, chronic gastrointestinal diseases or bowel resection.
* Cardiac disease.
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Inadequate bone marrow reserve or organ function.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2016-03-04 (Actual); Study Completion 2025-11-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- Australia (3):
  - Research Site, Kogarah
  - Research Site, Nedlands
  - Research Site, Woolloongabba
- China (14):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- South Korea (3):
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3720&filename=d5160c00017-csp-v3_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 22 June 2015, The study was open for enrollment at 31 study centres in China (24 sites), South Korea (4 sites), and Australia (3 sites)
Pre-assignment Details: 319 signed informed consent from 306 patients (13 patients were re-screened). Patients were assigned to treatment if they met all the inclusion and none of the exclusion criteria. 130 patients failed inclusion/exclusion criteria and 5 patients withdrew consent so were not eligible to be assigned treatment. Thus, 171 patients received treatment.
Period: Overall Study
Arm/Group | AZD9291
Started | 171
Completed | 46 (patients who terminated study due to study close out)
Not Completed | 125
Not completed — Death | 95
Not completed — Withdrawal by Subject | 27
Not completed — poor compliance after treatment discontinuation | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All patients enrolled who received at least 1 dose of study treatment.
Arm/Group | AZD9291
Number analyzed (Participants) | 171
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (10.81)
Age, Customized [Count of Participants; unit: Participants]
  <50 Years | 38
  >=50-<65 Years | 79
  >=65-<75 Years | 45
  >=75 Years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117
  Male | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 168
  White | 2
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: ORR According to RECIST 1.1 by Independent Review
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. ORR is the percentage of patients with at least 1 visit response of CR or PR (according to independent review) that was confirmed at least 4 weeks later, prior to progression or further anti-cancer therapy.
Time Frame: At baseline and every 6 weeks from time of first dose until objective disease progression,up to 24 months after Last Patient First Dose(LPFD)
Population: All patients who received at least 1 dose of study treatment and had measurable disease at baseline according to the independent review of baseline imaging data.
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | AZD9291
Number analyzed (Participants) | 166
% of participants | 62.0 [54.2 to 69.5]

2. Secondary Outcome: DoR According to RECIST 1.1 by Independent Review
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. DoR was defined as the time from the date of first documented response (CR or PR that was subsequently confirmed) until the date of documented progression (PD) or death in the absence of disease progression (by investigator assessment).
Time Frame: At baseline and every 6 weeks from time first dose until date of progression, up to 24 months after LPFD.
Population: All patients who received at least 1 dose of study treatment, had measurable disease at baseline according to the independent review of baseline imaging data and had confirmed response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AZD9291
Number analyzed (Participants) | 103
Months | 9.9 [8.3 to 12.9]

3. Secondary Outcome: DCR According to RECIST 1.1 by Independent Review
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions; Stable disease (SD): Neither sufficient shrinkage to qualify as a response nor sufficient growth to qualify as progression; Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. DCR is the percentage of patients with best response of CR, PR or SD (according to independent review), prior to progression (PD) or further anti-cancer therapy.
Time Frame: At baseline and every 6 weeks from time first dose until date of progression, up to 24 months after Last Patient First Dose(LPFD)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | AZD9291
Number analyzed (Participants) | 166
% of participants | 88.0 [82.0 to 92.5]

4. Secondary Outcome: Tumour Shrinkage According to RECIST 1.1 by Independent Review
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Tumour size was calculated as the sum of the longest diameters (SLD) of the Target Lesions. Tumour shrinkage is the best percentage change in tumour size from baseline using RECIST v1.1 tumour response.
Time Frame: At baseline and every 6 weeks from time of first dose until date of progression, up to 24 months after LPFD.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change from baseline in target lesion
Arm/Group | AZD9291
Number analyzed (Participants) | 166
% change from baseline in target lesion | -46.1 (28.40)

5. Secondary Outcome: PFS According to RECIST 1.1 by Independent Review
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. PFS is the time from date of first dose until the date of PD (by independent review) or death (by any cause in the absence of progression) regardless of whether the patient withdrew from AZD9291 therapy or received another anti-cancer therapy prior to progression. Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST 1.1 assessment.
Time Frame: At baseline and every 6 weeks from time of first dose until objective disease progression, up to 24 months after LPFD.
Population: All patients who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AZD9291
Number analyzed (Participants) | 171
Months | 9.7 [7.0 to 11.1]

6. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from first dose until death from any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Time Frame: From first dose to end of study or date of death from any cause, whichever comes first, assessed every 6 weeks up to approximately 95 OS events (about 55% maturity) have been observed out of all enrolled patients.
Population: All patients who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AZD9291
Number analyzed (Participants) | 171
Months | 23.2 [20.0 to 26.7]

ADVERSE EVENTS:
Time Frame: AEs were collected from time of signature of informed consent throughout the treatment period and including the 28-day safety follow-up after the last dose of the study treatment, approximately 33 months
Groups:
- AZD9291 80mg: Once daily tablet 80 mg
Arm/Group | AZD9291 80mg
All-Cause Mortality (participants affected / at risk) | 11/171
Serious Adverse Events (participants affected / at risk) | 42/171
Other Adverse Events (participants affected / at risk) | 163/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 80mg (N=171)
Sudden death (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Cataract (Eye disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (2)
Lung infection (Infections and infestations) | 3 (3)
Paronychia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 80mg (N=171)
Anaemia (Blood and lymphatic system disorders) | 25 (32)
Leukopenia (Blood and lymphatic system disorders) | 36 (90)
Neutropenia (Blood and lymphatic system disorders) | 20 (45)
Thrombocytopenia (Blood and lymphatic system disorders) | 25 (43)
Abdominal discomfort (Gastrointestinal disorders) | 12 (12)
Constipation (Gastrointestinal disorders) | 13 (18)
Diarrhoea (Gastrointestinal disorders) | 60 (186)
Mouth ulceration (Gastrointestinal disorders) | 11 (14)
Nausea (Gastrointestinal disorders) | 24 (32)
Vomiting (Gastrointestinal disorders) | 20 (23)
Asthenia (General disorders) | 10 (11)
Non-cardiac chest pain (General disorders) | 10 (13)
Pyrexia (General disorders) | 13 (26)
Hepatic function abnormal (Hepatobiliary disorders) | 9 (10)
Influenza (Infections and infestations) | 17 (28)
Paronychia (Infections and infestations) | 19 (26)
Upper respiratory tract infection (Infections and infestations) | 28 (53)
Urinary tract infection (Infections and infestations) | 17 (23)
Viral upper respiratory tract infection (Infections and infestations) | 24 (31)
Alanine aminotransferase increased (Investigations) | 13 (16)
Aspartate aminotransferase increased (Investigations) | 15 (23)
Blood creatinine increased (Investigations) | 14 (18)
Haemoglobin decreased (Investigations) | 12 (13)
Neutrophil count decreased (Investigations) | 19 (47)
Platelet count decreased (Investigations) | 31 (54)
Weight decreased (Investigations) | 9 (9)
White blood cell count decreased (Investigations) | 30 (68)
Decreased appetite (Metabolism and nutrition disorders) | 17 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (33)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (18)
Dizziness (Nervous system disorders) | 14 (19)
Headache (Nervous system disorders) | 15 (17)
Proteinuria (Renal and urinary disorders) | 9 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (58)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Dry skin (Skin and subcutaneous tissue disorders) | 26 (39)
Pruritus (Skin and subcutaneous tissue disorders) | 26 (51)
Rash (Skin and subcutaneous tissue disorders) | 18 (26)
Rash papular (Skin and subcutaneous tissue disorders) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days